CLINICAL TRIAL: NCT00005745
Title: Consequences and Correlates of Weight Fluctuations
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5006; R29HL057871 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-09

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Heart Diseases; Hypertension

SUMMARY:
To quantify the association between multiple intentional weight losses (i.e., weight fluctuations) and the development of hypertension and diabetes mellitus among 50,790 female nurses participating in the ongoing Nurses' Health Study II. In addition to assessing the consequences of weight fluctuations, their correlates and course were identified.

DETAILED DESCRIPTION:
BACKGROUND:

In the United States, approximately one third of adult women are trying to lose weight. Most weight losses are not sustained and in fact may be followed by gains of at least as much weight as was intentionally lost. It is unclear whether there are adverse outcomes associated with multiple intentional weight losses.

DESIGN NARRATIVE:

The prospective study addressed the impact of weight fluctuation on development of hypertension (HPT) and diabetes (DM) by following women who significantly fluctuated in weight compared to those who generally maintained a stable weight. The subject source was all participants between 1989 and 1993 in the Nurses Health Study II (NHS) who did not experience a full term pregnancy between 1989 and 1993 and who were free of HPT, DM and cancer in 1993. A random sample of each of two weight fluctuation classifications, >20 lbs. (3 or more times) and 10-19 lbs. (3 or more times) was identified. A control group of non-fluctuators was matched by age and body mass index strata. Baseline data consisted of information obtained from the 1993 NHS II follow-up along with supplemental questionnaires sent to study participants to elicit specific information on past and present weight gain/loss and intentionality of weight fluctuation. Prospective data came from follow-up questionnaires in 1995, 1997, and 1999. Hypertension and DM ascertainment were obtained from self-report in the questionnaire. This ascertainment method appeared quite adequate based on validity studies carried out on subsamples of this cohort.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-01; Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Field — Brigham and Women's Hospital

REFERENCES:
- [Background] Field AE, Wing RR, Manson JE, Spiegelman DL, Willett WC. Relationship of a large weight loss to long-term weight change among young and middle-aged US women. Int J Obes Relat Metab Disord. 2001 Aug;25(8):1113-21. doi: 10.1038/sj.ijo.0801643. PMID 11477495